CLINICAL TRIAL: NCT00638755
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Response Study to Evaluate the Effect of Nasal Carbon Dioxide on Nasal Congestion Via Acoustic Rhinometry in Subjects With Perennial Allergic Rhinitis
Brief Title: The Effect of Nasal Carbon Dioxide (CO2) on Nasal Congestion in Subjects With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capnia, Inc. (Industry)
Responsible Party: Kristen Yen- Associate Director, Clinical, Capnia, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C213
Record Dates: First submitted 2008-03-13; First posted 2008-03-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Allergic Rhinitis; Perennial Allergic Rhinitis; Allergies to perennial allergens; Allergies to perennial allergens (e.g. dog, cat, dust mites, etc.)
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): The following treatment sequence: A (Nasal Carbon Dioxide), B (Nasal Carbon Dioxide), C (Nasal Carbon Dioxide), D (placebo)
  Interventions: Drug: Nasal Carbon Dioxide
- 2 (Experimental): The following treatment sequence: B (Nasal Carbon Dioxide), C (Nasal Carbon Dioxide), D (placebo), A (Nasal Carbon Dioxide)
  Interventions: Drug: Nasal Carbon Dioxide
- 3 (Experimental): The following treatment sequence: C (Nasal Carbon Dioxide), D (placebo), A (Nasal Carbon Dioxide), B (Nasal Carbon Dioxide)
  Interventions: Drug: Nasal Carbon Dioxide
- 4 (Experimental): The following treatment sequence: D (placebo), A (Nasal Carbon Dioxide), B (Nasal Carbon Dioxide), C (Nasal Carbon Dioxide)
  Interventions: Drug: Nasal Carbon Dioxide

INTERVENTIONS:
Drug: Nasal Carbon Dioxide — Nasal Carbon Dioxide
  Arms: 1
Drug: Nasal Carbon Dioxide — Nasal Carbon Dioxide
  Arms: 2
Drug: Nasal Carbon Dioxide — Nasal Carbon Dioxide
  Arms: 3
Drug: Nasal Carbon Dioxide — Nasal Carbon Dioxide
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the effect of nasal CO2 on nasal congestion and other symptoms related to Perennial Allergic Rhinitis.

DETAILED DESCRIPTION:
A randomized study to evaluated the safety and effect of nasal carbon dioxide on nasal congestion using acoustic rhinometry in subjects with perennial allergic rhinitis. The acoustic rhinometry is an instrument that will be used to assess the levels of the nasal congestion in each subject. Approximately 20 men and women ages 19-65 years old who have a history consistent with perennial allergic rhinitis requiring pharmacology for at least 2 years and meet all other eligibility criteria will be enrolled in this study. There will be six (6) visits to the clinic. There will be a screening visit, four (4) treatment visits, and an end of study visit. A subject's participation in the study may last up to 58 days. There will be four different doses given in this study. Each subject will receive 3 different doses of the study drug and one dose of the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have a history consistent with minimal 2 year history of perennial allergic rhinitis requiring pharmacotherapy.
* Positive skin test to perennial allergens (e.g. cats, dogs, house dust mite, etc.)
* Females of childbearing potential must commit to using an acceptable method of birth control and have a negative pregnancy test

Exclusion Criteria:

* History of asthma (other than mild or intermittent)
* Clinically significant nasal disorders
* Acute or significant sinusitis or upper respiratory infection within 14 days of randomization
* Have an existing serious medical condition (such as severe emphysema, other respiratory diseases, heart disease, etc.) that precludes participation in the study
* Use of certain medication s prior to randomization and during study participation
* Participation in prior study with Nasal CO2
* Participation in another clinical study within 30 days of planned randomization date and for the duration of the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-07

PRIMARY OUTCOMES:
Determine the dose-related effects of CO2 on nasal congestion assessed by acoustic rhinometry. | Baseline, Post Treatment: 15 mins, 30 mins, 45 mins, 1 hour, 2 hours, 3 hours, 4 hours

SECONDARY OUTCOMES:
Change from baseline in olfactory test scores post-treatment | Baseline, Post Treatment: 1 hour & 3 hours
TNSS, TNNSS, and TSS comparisons at multiple timepoints | Baseline, Post Treatment: 15 mins, 30 mins, 45 mins, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 12 hours, 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Capnia Clinical Study Investigator, Principal Investigator — Capnia Investigative Site
Locations (1):
- Capnia Investigative Site, Omaha, Nebraska, United States